CLINICAL TRIAL: NCT01957280
Title: Phase 1, Open-label Study Assessing the Pharmacokinetics, Immunogenicity and Safety/Tolerability of Process 2 Patritumab in Patients With Advanced, Refractory Solid Tumors
Brief Title: Study to Assess Pharmacokinetics, Immunogenicity and Safety/Tolerability of Patritumab (U3-1287)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U31287-A-U105
Record Dates: First submitted 2013-06-12; First posted 2013-10-08 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Solid Tumors
Keywords: HER3
MeSH Terms: interventions — patritumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Process 2 patritumab (Experimental): Process 2 patritumab 18 mg/kg (loading dose) on Day 1 of Cycle 1 followed by Process 2 patritumab 9 mg/kg (maintenance dose) once every 21 days starting on Day 1 of Cycle 2 through Cycle 5.
  Interventions: Drug: patritumab

INTERVENTIONS:
Drug: patritumab
  Other Names: U3-1287

SUMMARY:
The purpose of this study is to assess the PK, safety, and tolerability of patritumab produced by a new manufacturing process (denoted as "Process 2 patritumab"). The data from this study will allow Process 2 patritumab to be compared to Process 1 patritumab to allow for any dose adjustments, if needed, and to bridge data from studies previously conducted with Process 1 patritumab to studies to be conducted with Process 2 patritumab. The hypothesis for this study is that the pharmacokinetics of Process 2 patritumab will be comparable to those of Process 1 patritumab.

DETAILED DESCRIPTION:
Process 2 patritumab will be administered intravenously as a single, loading dose of 18 mg/kg over approximately 60 minutes at Cycle 1 Day 1 followed by 9 mg/kg administered every 21 days as a maintenance dose starting at Cycle 2 Day 1. This study will be conducted in 2 phases: a main study and an extension phase. The PK profile of Process 2 patritumab will be compared to historical data for Process 1 patritumab. Specifically, the PK parameters (AUC0-21d and Cmax as primary endpoints) for Process 2 patritumab 18 mg/kg (loading dose) will be compared to the PK parameters of Process 1 patritumab 18 mg/kg. Process 2 patritumab serum concentrations will be compared to Process 1 patritumab serum concentrations collected in the Phase 1 and Phase 2 studies by population PK methods and will be reported separately.

ELIGIBILITY:
Inclusion Criteria:

* Must have a pathologically documented advanced solid tumor that is refractory to standard treatment, for which no standard therapy is available, or for which the subject refuses standard therapy.
* Must have a tumor type that is known to express HER3. These tumors include breast, lung, prostate, ovarian, cervical, endometrial, gastric, pancreatic, bladder, head and neck, liver, colon, and esophageal cancer. Other tumors will be considered based on emerging HER3 expression data.
* Must be competent and able to comprehend, sign, and date an IRB-approved ICF (including HIPAA authorization, if applicable) before performance of any study-specific procedures or tests.
* Must have an ECOG performance status of ≤ 2
* Women must be one of the following:

  1. Postmenopausal (having had no menstrual period for a minimum of 12 months) or surgically sterile, or
  2. If of childbearing potential, must have been willing to use maximally effective birth control during the period of therapy and use contraception for 6 months following the last investigational drug infusion and must have had a negative urine or serum pregnancy test upon entry into the study.
* Men must be surgically sterile or willing to use a double-barrier contraception method upon enrollment, during the course of the study, and for 6 months following the last investigational drug infusion.
* Have hematological function, as follows:6. Men

  * Absolute neutrophil count of ≥ 1.5 × 109/L
  * Platelet count ≥ 100 × 109/L
  * Hemoglobin ≥ 9 g/dL
* Have renal function, as follows:

  * Calculated creatinine clearance rate (CrCl) ≥ 60 mL/minute using the modified Cockcroft-Gault equation or serum creatinine ≤ 1.5 × ULN.
* Have hepatic function, as follows:

  * AST ≤ 2.5 × ULN (if liver metastases are present, < 5 × ULN)
  * ALT ≤ 2.5 × ULN (if liver metastases are present, < 5 × ULN)
  * Alkaline phosphatase ≤ 2.5 × ULN (if bone or liver metastases are present, < 5 × ULN)
  * Bilirubin ≤ 1.5 × ULN
  * Prothrombin time (PT) or partial thromboplastin time (PTT) ≤ 1.5 × ULN

Exclusion Criteria:

* Have a history of lymphoma, leukemia, or other hematopoietic malignancy.
* Have Have autologous or allogeneic stem cell transplant.
* Have any comorbid medical condition that would increase the risk of toxicity in the opinion of the investigator or sponsor.
* Have untreated or symptomatic brain metastasis.
* Have unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE Version 4.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia. Subjects with irreversible Grade 2 toxicity may be eligible as per discretion of the investigator and sponsor (e.g., Grade 2 chemotherapy-induced neuropathy).
* Have uncontrolled hypertension (diastolic blood pressure > 100 mmHg or systolic blood pressure > 140 mmHg). It is permissible for the subject to receive treatment with antihypertensive medication to maintain blood pressure within the required parameters.
* Have clinically significant ECG changes that obscure the ability to assess the RR, PR, QT, QT interval corrected for heart rate (QTc), and QRS interval. Subjects with left bundle branch block, atrial fibrillation and use of cardiac pacemaker specifically will be excluded.
* Have ascites or pleural effusion requiring chronic medical intervention.
* Have a history of bleeding diathesis.
* Have had a myocardial infarction within 1 year before enrollment, symptomatic CHF (New York Heart Association > Class II;), unstable angina, or unstable cardiac arrhythmia requiring medication.
* Use of amiodarone within 6 months prior to enrollment.
* Concurrent use of antiarrhythmic medications with the exception of beta blockers for treatment of hypertension.
* Subjects who are receiving drugs that may affect QTc (e.g., quinidine or moxifloxacin).
* QTc interval > 450 msec on the average of the triplicate readings by Friderica's formula on 2 successive screening measurements (second measurement is required if first measurement is > 450 msec).
* Have a LVEF < 50%.
* Have anthracycline exposure greater than 360 mg/m2.
* Have a history of chronic hepatitis or known active infection with hepatitis B virus or hepatitis C virus.
* Personal or family history of long-QT syndrome.
* Have known infection with or a history of testing positive for human immunodeficiency virus (HIV).
* Had treatment with anticancer therapy (6 weeks for nitrosoureas and mitomycin C chemotherapies and 2 weeks for small molecule tyrosine kinase inhibitors), antibody therapy, retinoid therapy, or hormonal therapy within 4 weeks before study Day 1. Prior and concurrent use of hormone replacement therapy or the use of gonadotropin releasing hormone modulators for prostate cancer is permitted.
* Had therapeutic or palliative radiation therapy within 4 weeks before enrollment (in addition, he/she must have had resolution of any significant AEs from radiation therapy at least 2 weeks before enrollment).
* Have concurrent or previous (within 1 week of study Day 1) anticoagulation therapy, except low-dose warfarin (≤ 2 mg/day) or low-dose, low-molecular weight heparin for prophylaxis against central venous catheter thrombosis or deep vein thrombosis.
* Have participated in clinical drug trials within 4 weeks before enrollment.
* Have had major surgery within 4 weeks before enrollment.
* Is currently participating in other investigational procedures.
* Has any disorder that compromised the ability of the subject to give written informed consent and/or comply with study procedures.
* Has known sensitivity to any of the products to be administered during dosing or known allergy to the excipients or investigational drugs.
* Has active infection within 2 weeks before enrollment unless there was a discussion with the sponsor and an agreement was reached that the recent infection would not affect the subject's participation in the study.
* Has previously received an anti-HER3 targeted antibody, including patritumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
AUC (0-21 day) of Patritumab | 5 Cycles, each of which lasts 21 Days
  AUC (0-21 day) of patritumab obtained after a single infusion of Process 2 patritumab 18 mg/kg (loading dose)
Cmax of Patritumab | 5 Cycles, each of which lasts 21 Days
  Cmax of patritumab obtained after a single infusion of Process 2 patritumab 18 mg/kg (loading dose)

SECONDARY OUTCOMES:
volume of distribution [Vz] | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameters volume of distribution [Vz]
Safety and Tolerability of Process 2 patritumab - (electrocardiograms [ECG) | 5 Cycles, each of which lasts 21 Days
  To assess the safety and tolerability of Process 2 patritumab (electrocardiograms [ECG)
Antibody Formation | 5 Cycles, each of which lasts 21 Days
  To characterize the formation of antibodies to patritumab human antihuman antibodies (HAHA) after infusion of Process 2 patritumab
Concentration patritumab at 504 hours | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameter concentration of patritumab at 504h [C504]
AUC to infinity [AUC0-inf] | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameters AUC to infinity [AUC0-inf]
time to Cmax (Tmax) | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameters time to Cmax (Tmax)
concentration at the end of infusion (Ceoi) | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameters concentration at the end of infusion (Ceoi)
terminal elimination half-life (t 1/2) | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameters terminal elimination half-life (t 1/2)
clearance (CL) | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameters clearance (CL)
trough concentration (Ctrough) | 5 Cycles, each of which lasts 21 Days
  To assess the secondary PK parameters trough concentration (Ctrough)
echocardiograms/multi-gated acquisition [MUGA] scans of Process 2 patritumab | 5 Cycles, each of which lasts 21 Days
  To assess the safety and tolerability of Process 2 patritumab echocardiograms/multi-gated acquisition [MUGA] scans
adverse events [AEs] of Process 2 patritumab | 5 Cycles, each of which lasts 21 Days
  To assess the safety and tolerability of Process 2 patritumab adverse events [AEs] of Process 2 patritumab

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tampa, Florida
  - Oklahoma City, Oklahoma
  - San Antonio, Texas